CLINICAL TRIAL: NCT01539083
Title: An Open-label, Randomised Trial of Bortezomib Consolidation (With Thalidomide and Prednisolone) Vs Thalidomide and Prednisolone Alone in Previously Untreated Subjects With Multiple Myeloma After Receiving Bortezomib, Cyclophosphamide, Dexamethasone (VCD) Induction and Autologous Stem Cell Transplant
Brief Title: Velcade (Bortezomib) Consolidation After Transplant
Acronym: VCAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018751; 26866138-MMY-2073 (Other: Janssen Asia-Pacific Medical Affairs)
Record Dates: First submitted 2011-11-23; First posted 2012-02-27 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; VELCADE; Consolidation therapy; Subcutaneous; Thalidomide; Prednisolone; Autologous stem cell transplant (ASCT); VELCADE, cyclophosphamide, dexamethasone (VCD) induction therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Bortezomib; Cyclophosphamide; Dexamethasone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bortezomib + Cyclophosphamide + Dexamethasone [VCD Induction] (Experimental): Bortezomib (Velcade) 1.3 milligram per square meter (mg/m^2) subcutaneously (SC) on Days 1, 4, 8, and 11; cyclophosphamide 300 mg/m^2 orally on Days 1, 8, and 15; and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11, and 12 in three 21-day treatment cycles. Participants who completed induction phase entered into the consolidation treatment phase.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone
- Thalidomide + Prednisolone [TP Consolidation] (Experimental): Thalidomide 100 mg orally, once daily until disease progression (up to maximum of 12 months) and prednisolone 50 mg orally, on every alternate day until disease progression.
  Interventions: Drug: Thalidomide; Drug: Prednisolone
- Bortezomib + Thalidomide + Prednisolone [VTP Consolidation] (Experimental): Bortezomib 1.3 mg/m^2 SC every 2 weeks for 32 weeks in addition to thalidomide 100 mg orally, once daily for a maximum of 12 months or until disease progression and prednisolone 50 mg orally, on every alternate day until disease progression.
  Interventions: Drug: Thalidomide; Drug: Bortezomib; Drug: Prednisolone

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 100 mg tablet, orally.
  Arms: Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]; Thalidomide + Prednisolone [TP Consolidation]
Drug: Bortezomib — Bortezomib 1.3 milligram per square meter (mg/m^2) solution for injection subcutaneously (SC).
  Arms: Bortezomib + Cyclophosphamide + Dexamethasone [VCD Induction]; Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Drug: Cyclophosphamide — Cyclophosphamide 300 mg/m^2 orally.
  Arms: Bortezomib + Cyclophosphamide + Dexamethasone [VCD Induction]
Drug: Dexamethasone — Dexamethasone 20 mg orally.
  Arms: Bortezomib + Cyclophosphamide + Dexamethasone [VCD Induction]
Drug: Prednisolone — Prednisolone 50 mg orally.
  Arms: Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]; Thalidomide + Prednisolone [TP Consolidation]

SUMMARY:
The purpose of this study is to determine if bortezomib when added to consolidation treatment with thalidomide and prednisolone leads to an improved response in patients with multiple myeloma who have undergone autologous stem cell transplant and initial treatment with bortezomib, cyclophosphamide, and dexamethasone.

DETAILED DESCRIPTION:
This is an open-label (patients will know the identity of study treatments), randomized (patients will be assigned by chance to different treatments) study of bortezomib administered as consolidation therapy (therapy given once a remission is achieved) with thalidomide and prednisolone versus thalidomide and prednisolone alone in previously untreated patients with multiple myeloma. Multiple myeloma is a cancer of your plasma cells, a type of white blood cell present in your bone marrow. Patients in this study will receive initial therapy with bortezomib, cyclophosphamide, and dexamethasone (referred to as VCD induction therapy) and will undergo autologous stem cell transplant (ASCT) (a procedure where patients receive an infusion of immature blood cells [stem cells] from their own body to replenish the body's supply of healthy blood-forming cells) before randomization to one of two treatments: Treatment A (thalidomide for up to 12 months or until disease progression and prednisolone on alternate days continued indefinitely or until disease progression) or Treatment B (bortezomib for 32 weeks in addition to thalidomide up to 12 months or until disease progression and prednisolone on alternate days, continued indefinitely or until disease progression.

Throughout the study, the patient's response to therapy will be assessed according to protocol-defined efficacy evaluations and by implementing defined disease response criteria (International Myeloma Working Group [IMWG] criteria). Safety will be evaluated throughout the study. Follow up for progression-free survival (PFS) and overall survival (OS) will be conducted from time of randomization to 3 years post-randomization.

Two interim analyses are planned. The final analysis will be conducted after all patients have completed 12-month consolidation treatment phase or discontinued. The primary endpoint of number and percent of patients with complete response and very good partial response defined by IMWG criteria for multiple myeloma will be examined in the interim and final analyses after approximately 12 months of consolidation therapy. At the completion of the study, updated analyses of PFS and OS will be performed.

ELIGIBILITY:
Inclusion criteria:

* Previously diagnosed with multiple myeloma based on international myeloma working group (IMWG) criteria.and meet all of the following; Serum M-protein greater than or equal to (>=) 1 gram per deciliter (g/dL) (>=10 gram per liter); Urine M-protein >=200 milligram (mg) per 24 hour and Serum Free Light chain (FLC) assay: Involved FLC Level >=10 mg/dL (>=100 mg/L) provided serum FLC ratio is normal
* Meet the pretreatment laboratory criteria as specified in the study protocol at and within 21 days before baseline (Day 1 of Cycle 1, before bortezomib administration for induction).
* Have ECOG status 0-2.
* Men and women must practice an appropriate method of birth control as specified in the study protocol from signing of the informed consent form though to the 12-month visit/early termination visit.

Exclusion criteria:

* Has previously received treatment for multiple myeloma (including prior therapy with radiation or pulsed dexamethasone) as specified in the study protocol.
* Has a history of any other malignancy within 5 years before enrolment as specified in the study protocol.
* Has had major surgery as specified in the study protocol within 30 days before enrolment.
* Had a myocardial infarction within 6 months of enrolment or has New York Heart Association (NYHA) Class III or IV heart failure (or other clinically significant cardiac medical history as specified in the study protocol).
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Asia-Pacific Medical Affairs Clinical Trial, Study Director — Janssen Asia-Pacific Medical Affairs
Locations (23):
- Australia (15):
  - Adelaide
  - Camperdown
  - Geelong
  - Greenslopes
  - Heidelberg
  - Herston
  - Malvern
  - Melbourne
  - Nedlands
  - Newcastle
  - Prahran
  - Sydney
  - Westmead
  - Woodville South
  - Woolloongabba
- China (4):
  - Beijing
  - Guangzhou
  - Shanghai
  - Tianjin
- South Korea (4):
  - Busan
  - Daegu
  - Jeollanam-do
  - Ulsan

REFERENCES:
- [Derived] Horvath N, Spencer A, Kenealy M, Joshua D, Campbell PJ, Lee JJ, Hou J, Qiu L, Kalff A, Khong T, Londhe A, Siggins S, van Kooten Losio M, Eisbacher M, Prince HM. Phase 3 study of subcutaneous bortezomib, thalidomide, and prednisolone consolidation after subcutaneous bortezomib-based induction and autologous stem cell transplantation in patients with previously untreated multiple myeloma: the VCAT study. Leuk Lymphoma. 2019 Sep;60(9):2122-2133. doi: 10.1080/10428194.2019.1579322. Epub 2019 Feb 19. PMID 30777794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 treatment phases: induction and consolidation. Participants who completed the induction phase were randomized to enter in the consolidation treatment phase.
Groups:
- Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction): Participants received bortezomib (Velcade) 1.3 milligram per square meter (mg/m^2) subcutaneously (SC) on Days 1, 4, 8, and 11; cyclophosphamide 300 mg/m^2 orally on Days 1, 8, and 15; and dexamethasone 20 milligram (mg) orally on Days 1, 2, 4, 5, 8, 9, 11, and 12 in three 21-day treatment cycles. Participants who completed induction phase entered into the consolidation treatment phase.
- Thalidomide + Prednisolone (TP Consolidation): Participants who completed induction phase entered in the consolidated treatment phase and received thalidomide 100 mg orally, once daily until disease progression (up to maximum of 12 months) and prednisolone 50 mg orally, on every alternate day until disease progression.
- Bortezomib + Thalidomide + Prednisolone (VTP Consolidation): Participants who completed induction phase entered in the consolidated treatment phase and received bortezomib 1.3 mg/m^2 SC every 2 weeks for 32 weeks in addition to thalidomide 100 mg orally, once daily for a maximum of 12 months or until disease progression and prednisolone 50 mg orally, on every alternate day until disease progression.
Period: Before Randomization (VCD Induction)
Arm/Group | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction) | Thalidomide + Prednisolone (TP Consolidation) | Bortezomib + Thalidomide + Prednisolone (VTP Consolidation)
Started | 256 | 0 | 0
Treated | 254 | 0 | 0
Completed | 203 | 0 | 0
Not Completed | 53 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0
Not completed — Death | 6 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Physician Decision | 14 | 0 | 0
Not completed — Progressive Disease | 8 | 0 | 0
Not completed — Other | 5 | 0 | 0
Period: After Randomization (TP and VTP)
Arm/Group | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction) | Thalidomide + Prednisolone (TP Consolidation) | Bortezomib + Thalidomide + Prednisolone (VTP Consolidation)
Started | 0 | 100 (Participants who completed induction phase were randomized for the consolidated treatment.) | 103 (Participants who completed induction phase were randomized for the consolidation treatment phase.)
Safety Population | 0 | 99 (One participant was randomized but not treated. Hence, was not included in safety population.) | 103
Completed | 0 | 79 | 80
Not Completed | 0 | 21 | 23
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Other | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 5 | 4
Not completed — Progressive Disease | 0 | 6 | 3
Not completed — Death | 0 | 6 | 11

BASELINE CHARACTERISTICS:
Population: Baseline population was defined as all enrolled participants who received at least 1 non-zero dose of any study drug in the induction phase.
Arm/Group | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction)
Number analyzed (Participants) | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 145
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 207
  China | 17
  Republic of Korea | 30

OUTCOME MEASURES:

1. Primary Outcome: Consolidation Phase: Percentage of Participants With Complete Response (CR) and Very Good Partial Response (VGPR) at Month 12
Description: CR as per IMWG criteria is defined as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and less than (<) 5 percent plasma cells in bone marrow. VGPR as per IMWG criteria is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90 percent or greater reduction in serum M-protein plus urine M-protein level <100 milligram (mg) per 24 hours.
Time Frame: Month 12
Population: All response-evaluable-randomized analysis set was defined as all participants in the response-evaluable-induction set (all participants who received at least 1 dose of study medication in the induction phase and had measurable disease at baseline) who were randomized to receive consolidation treatment.
Measure: Number; unit: percentage of participants
Groups:
- Thalidomide + Prednisolone [TP Consolidation]: Participants who completed induction phase entered in the consolidated treatment phase and received thalidomide 100 mg orally, once daily until disease progression (up to maximum of 12 months) and prednisolone 50 mg orally, on every alternate day until disease progression.
- Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]: Participants who completed induction phase entered in the consolidated treatment phase and received bortezomib 1.3 mg/m^2 SC every 2 weeks for 32 weeks in addition to thalidomide 100 mg orally, once daily for a maximum of 12 months or until disease progression and prednisolone 50 mg orally, on every alternate day until disease progression.
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 96 | 98
percentage of participants | 81.3 | 92.9

2. Secondary Outcome: Consolidation Phase: Percentage of Participants With Complete Response (CR) at Months 3, 6, 9 and 12
Description: CR as per IMWG criteria is negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and <5 percent plasma cells in bone marrow.
Time Frame: Months 3, 6, 9 and 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 96 | 98
percentage of participants
  Month 3 | 36.5 | 36.7
  Month 6 | 44.8 | 44.9
  Month 9 | 49.0 | 52.0
  Month 12 | 51.0 | 53.1

3. Secondary Outcome: Consolidation Phase: Percentage of Participants With Stringent Complete Response (sCR) at Months 3, 6, 9 and 12
Description: sCR as per IMWG criteria is CR plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow. CR is negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and <5 percent plasma cells in bone marrow.
Time Frame: Months 3, 6, 9 and 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 96 | 98
percentage of participants
  Month 3 | 20.8 | 23.5
  Month 6 | 27.1 | 28.6
  Month 9 | 26.0 | 30.6
  Month 12 | 26.0 | 28.6

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, calculated as the time between randomization to disease progression or death (regardless of cause), whichever occurred first. Progressive disease as per IMWG criteria: increase of >= 25 percent from lowest response level in Serum M-component and/or (the absolute increase must be >=0.5 gram per deciliter [g/dL]) Urine M-component and/or (the absolute increase must be >=200 mg/24 hour. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels. The absolute increase must be >10 mg/dL. Bone marrow plasma cell percentage: the absolute percent must be >=10 percent. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65 millimole per liter (mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: Baseline until progressive disease (up to 5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 96 | 98
months | 22.05 [18.46 to 25.49] | 22.51 [18.56 to 24.15]

5. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS, defined as the duration from the start of CR to the time of relapse from CR. DFS applied only to participants in CR. CR as per IMWG criteria is negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and <5 percent plasma cells in bone marrow. Relapse from CR: reappearance of serum or urine M-protein by immunofixation or electrophoresis; development of >= 5 percent plasma cells in the bone marrow; appearance of any other sign of progression (ie, new plasmacytoma, lytic bone lesion, or hypercalcaemia).
Time Frame: Up to 5 years
Population: Response-evaluable-randomized analysis set defined as all participants in the response-evaluable-induction set (who received at least 1 dose of study medication;had measurable disease at baseline) who were randomized to receive consolidation treatment. Here, 'N' (number of participants analyzed) signifies the participants who had complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 56 | 62
months | 18.53 [11.24 to 23.36] | 13.37 [10.18 to 20.96]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between randomization and death. Death of a participant regardless of the cause was considered as an event.
Time Frame: Up to 5 years
Population: All randomized analysis set was defined as participants in the all enrolled set (all participants with a non-missing informed consent date and were not screen failures) who were randomized to receive consolidation treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 100 | 103
months | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events.

7. Secondary Outcome: Consolidation Phase: Change From Baseline in AQOL-6D Scores at the End of the Consolidation Phase
Description: The assessment of quality of life-6D (AQoL-6D) is a multi-attribute health-related quality of life instrument (QoL). It comprises dimension scores for independent living, relationships, mental health, coping, pain, senses, and utility score for AQol-6D. Each scale ranges between 1 (best QoL) and -0.04 (worst possible QoL).
Time Frame: Baseline, Month 12
Population: All treated randomized analysis set was defined as participants in the all enrolled set (participants with non-missing informed consent date,not screen failures) received at least 1 dose of any study drug and randomized to receive consolidation treatment. Here, 'N'(number of participants analyzed) participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 83 | 86
units on a scale
  Independent Living | 0.15 (0.335) | 0.14 (0.397)
  Relationships | 0.06 (0.300) | 0.05 (0.296)
  Mental Health | 0.18 (0.319) | 0.18 (0.270)
  Coping | 0.08 (0.278) | 0.05 (0.237)
  Pain | 0.20 (0.373) | 0.20 (0.395)
  Senses | 0.03 (0.140) | 0.00 (0.137)
  AQoL-6D Utility score | 0.11 (0.216) | 0.11 (0.213)

8. Secondary Outcome: Consolidation Phase: Change From Baseline in FACT/GOG-NTX Total Score at the End of the Consolidation Phase
Description: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) consists of 10 items and evaluates symptoms and concerns associated specifically with chemotherapy-induced neuropathy. 1 FACT/GOG-NTX total score has a range of 0 to 108 with a higher score indicating better quality of life.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thalidomide + Prednisolone [TP Consolidation] | Bortezomib + Thalidomide + Prednisolone [VTP Consolidation]
Number analyzed (Participants) | 83 | 86
units on a scale | 2.9 (19.68) | 1.0 (19.69)

ADVERSE EVENTS:
Description: Safety population included all participants in the induction and consolidation phase who received at least 1 dose of study drug.
Arm/Group | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction) | Thalidomide + Prednisolone (TP Consolidation) | Bortezomib + Thalidomide + Prednisolone (VTP Consolidation)
Serious Adverse Events (participants affected / at risk) | 88/254 | 22/99 | 28/103
Other Adverse Events (participants affected / at risk) | 233/254 | 95/99 | 96/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction) (N=254) | Thalidomide + Prednisolone (TP Consolidation) (N=99) | Bortezomib + Thalidomide + Prednisolone (VTP Consolidation) (N=103)
Febrile Neutropenia (Blood and lymphatic system disorders) | 11 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Oesophageal Spasm (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Adverse Drug Reaction (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 12 | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1
Bacillus Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 2
Herpes Zoster Disseminated (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 2 | 0
Localised Infection (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 1 | 2
Lung Infection (Infections and infestations) | 2 | 0 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 6 | 7
Pneumonia Influenzal (Infections and infestations) | 0 | 0 | 1
Pneumonia Primary Atypical (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 4 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cytomegalovirus Test Positive (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Embolic Stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diaphragmatic Paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Embolism Venous (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Cyclophosphamide + Dexamethasone (VCD Induction) (N=254) | Thalidomide + Prednisolone (TP Consolidation) (N=99) | Bortezomib + Thalidomide + Prednisolone (VTP Consolidation) (N=103)
Anaemia (Blood and lymphatic system disorders) | 25 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 17 | 0 | 5
Tinnitus (Ear and labyrinth disorders) | 2 | 5 | 8
Cushingoid (Endocrine disorders) | 0 | 6 | 3
Vision Blurred (Eye disorders) | 8 | 8 | 7
Visual Impairment (Eye disorders) | 1 | 6 | 2
Constipation (Gastrointestinal disorders) | 91 | 38 | 29
Diarrhoea (Gastrointestinal disorders) | 32 | 14 | 15
Dry Mouth (Gastrointestinal disorders) | 6 | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 14 | 3 | 1
Nausea (Gastrointestinal disorders) | 82 | 10 | 12
Vomiting (Gastrointestinal disorders) | 32 | 7 | 3
Chest Pain (General disorders) | 9 | 5 | 2
Fatigue (General disorders) | 61 | 18 | 16
Injection Site Rash (General disorders) | 14 | 0 | 1
Injection Site Reaction (General disorders) | 19 | 0 | 7
Oedema Peripheral (General disorders) | 44 | 15 | 16
Herpes Zoster (Infections and infestations) | 8 | 10 | 5
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 5 | 6
Nasopharyngitis (Infections and infestations) | 5 | 5 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 29 | 32 | 39
Contusion (Injury, poisoning and procedural complications) | 4 | 6 | 3
Weight Increased (Investigations) | 7 | 26 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 19 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 9 | 12
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 9 | 11
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 14 | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 | 7 | 7
Dizziness (Nervous system disorders) | 23 | 7 | 7
Dysgeusia (Nervous system disorders) | 21 | 2 | 0
Headache (Nervous system disorders) | 21 | 8 | 5
Hypoaesthesia (Nervous system disorders) | 10 | 6 | 6
Lethargy (Nervous system disorders) | 16 | 3 | 6
Neuralgia (Nervous system disorders) | 19 | 14 | 16
Neuropathy Peripheral (Nervous system disorders) | 34 | 24 | 30
Paraesthesia (Nervous system disorders) | 11 | 7 | 9
Peripheral Sensory Neuropathy (Nervous system disorders) | 62 | 38 | 38
Tremor (Nervous system disorders) | 12 | 11 | 11
Insomnia (Psychiatric disorders) | 56 | 22 | 13
Mood Altered (Psychiatric disorders) | 9 | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 6
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 22 | 7 | 10
Hypertension (Vascular disorders) | 2 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.